CLINICAL TRIAL: NCT01080638
Title: Intracoronary Bolus Only Compared With Intravenous Bolus and 12-hours Infusion of Abciximab in Non-ST Elevation Myocardial Infarction.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other)
Responsible Party: Hyo-Soo Kim/ Prof, Director of Cardiac Catheterization Laboratory & Coronary Intervention of Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-0906-046-283
Record Dates: First submitted 2010-02-16; First posted 2010-03-04 (Estimated); Last update posted 2010-03-04 (Estimated); Status verified 2010-03

CONDITIONS: Myocardial Infarction; Angioplasty
Keywords: abciximab; Myocardial Infarction; angioplasty; Platelet
MeSH Terms: conditions — Myocardial Infarction | interventions — Abciximab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Abciximab IC bolus (Experimental): After CAG, For patients with undergoing percutaneous coronary intervention, intracoronary only or intravenous bolus abciximab(0.25mg/kg body weight) administration with intravenous bolus group has subsequent 12-hours continuous infusion at a dose 0.125ug/kg per minute (maximum: 10ug/min)
  Interventions: Drug: glycoprotein IIb/IIIa inhibitor (abciximab)
- Abciximab IV bolus and 12hr continuous (Active Comparator)
  Interventions: Drug: glycoprotein IIb/IIIa inhibitor (abciximab)

INTERVENTIONS:
Drug: glycoprotein IIb/IIIa inhibitor (abciximab) — patients intracoronary bolus only group and intravenous bolus and 12-hours continuous infusion group bolus:0.25mg/kg body weight,continus 12hrs-0.125ug/kg per minute(maximum: 10ug/min)

SUMMARY:
Intracoronary bolus Abciximab single is non-inferior to intravenous and continuous 12- hours infusion in the size reduction of infarction on cardiac magnetic resonance in Non-ST elevation Myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* non-ST segment elevation acute myocardial infarction
* within 48 hours presence of chest pain
* Troponin-T or I positive before CAG
* First myocardial infarction
* will be performed coronary angioplasty

Exclusion Criteria:

* under 18 years of age,80 years or older
* Bleeding tendency
* History of major surgery within 4 weeks
* Major stroke within 2 years
* Thrombocytopenia (<120,000 / uL)
* Cardiogenic shock
* Known allergy to aspirin, heparin, or abciximab
* Contraindication of MRI at study entry (implanted pacemakers, defibrillators, intracranial metallic implants etc)
* Chronic atrial fibrillation
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
In cardiac MRI- infarct size (total late enhancement volume at day 3-7) | day 3~7 after percutaneous coronary intervention
  MRI: magnetic resonance image

SECONDARY OUTCOMES:
in-hospital and after 1-months:the major adverse cardiovascular events : death, myocardial infarction, hospitalization for heart failure, myocardial ischemia, etc. | 1 month
b. major bleeding : Hemoglobin 4 or more reduction, 2-unit If you need more than two RBC transfusions, intracranial or retroperitoneal bleeding, urgent operation for bleeding complication. | 1 month
  RBC: red blood cell
TIMI III flow count /myocardial blush score after PCI | 1 day
  TIMI: thrombolysis in myocardial infarction PCI: percutaneous coronary intervention
At cardiac MRI : LV ejection fraction,LV end-systolic volume,LV end diastolic volume,regional wall motion score index | 1 week
  LV: left ventricle
Discharge, 1- month after comparing NT-proBNP | 1 month
  NT-proBNP : N-terminal pro-B-Type natriuretic peptide

CONTACTS AND LOCATIONS:
Overall Officials: Hyun-Jae Kang, Prof, Study Director — Assistant professor, Cardiology, Department of internal medicine,Seoul National University Hospital
Locations (1):
- Department of Internal Medicine, Cardiovascular Center, Seoul National University Hospital, Seoul, South Korea